CLINICAL TRIAL: NCT03172962
Title: Effect of Strength Training for Chronic Low Back Pain Patients: Randomized Clinical Trial
Brief Title: Effect of Strength Training for Chronic Low Back Pain Patients (IRMA20)
Acronym: IRMA20
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre for the Working Environment, Denmark (Other Government)
Collaborators: University of Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRMA20
Record Dates: First submitted 2017-05-30; First posted 2017-06-01 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Musculoskeletal Pain; Low Back Pain
MeSH Terms: conditions — Musculoskeletal Pain; Low Back Pain | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strength training (Experimental): Specific strength training exercises for the lumbar and abdominal muscles for 8 weeks
  Interventions: Behavioral: Strength training; Behavioral: Usual care (control)
- Usual care (control) (Active Comparator): Will receive the usual care at the hospital
  Interventions: Behavioral: Usual care (control)

INTERVENTIONS:
Behavioral: Strength training — Specific strength training exercises for the lumbar and abdominal muscles for 8 weeks
  Arms: Strength training
Behavioral: Usual care (control) — Will receive the usual care at the hospital

SUMMARY:
Low back pain (LBP) is common in the population and has great socioeconomic consequences for societies across Europe and the United States. About a third of working-age adults have frequent LBP, and for about 10% the pain becomes chronic with consequences for work and leisure activities. A Cochrane review from April 2017 concluded that physical exercise is an intervention with few adverse events and positive outcomes on pain and function in adults with chronic pain. However, when scrutinizing the specific studies of the review there are large differences in adherence to the exercise interventions and consequently in the results obtained. Thus, there is a need for simple exercises that the patients can easily adhere to.

ELIGIBILITY:
Inclusion Criteria:

* Non-specific Chronic low back pain patient (more than 3 months) at the hospital Arnau de Vilanova

Exclusion Criteria:

* Spine surgery
* neurologic or psyquiatric disorders
* Low back traumastism
* Recent participation in a similar training program

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Low back pain intensity | change from baseline to 8-week follow-up
  Low back pain intensity (VAS 0-10)
Back pain recurrence | 1 to 100 days, beginning from the last day of termination of the 8-week intervention
  number of episodes with back pain recurrence after termination of the intervention

SECONDARY OUTCOMES:
Roland-Morris disability | change from baseline to 8-week follow-up
  The Roland-Morris disability questionnaire
Muscle endurance | change from baseline to 8-week follow-up
  The Biering-Sørensen test
Use of analgesics | change from baseline to 8-week follow-up
  Number of days using analgesic within the last week
Handgrip strength | change from baseline to 8-week follow-up
  Maximal force (kg) in handgrip
Pain sites | change from baseline to 8-week follow-up
  Number of pain sites

CONTACTS AND LOCATIONS:
Overall Officials: Joaquin Calatayud, PhD, Principal Investigator — University of Valencia
Locations (1):
- Primary care center of Lliria, Llíria, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided